CLINICAL TRIAL: NCT03858569
Title: Effect of Uterine Massage on Postpartum Hemorrhage After Vaginal Delivery
Brief Title: Uterine Massage After Vaginal Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/11/42
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): 10 units of oxytocin will be given intramuscularly immediately after delivery of the fetus
  Interventions: Procedure: active management of third stage of labor
- Oxytocin plus uterine massage (Active Comparator): 10 units of oxytocin will be given intramuscularly immediately after delivery of the fetus and transabdominal uterine massage will be performed.
  Interventions: Procedure: active management of third stage of labor

INTERVENTIONS:
Procedure: active management of third stage of labor — Active management of the third stage of the labor will be done administering oxytocin and cord traction.

SUMMARY:
The participants will be randomized into an oxytocin plus uterine massage group and an oxytocin-only group in the third stage of the labor. Women allocated to the uterine massage group will be provided with trans-abdominal uterine massage starting promptly after delivery of the fetus until delivery of the placenta. The amount of postpartum hemorrhage and placental delivery time will be recorded and compared between the groups.

DETAILED DESCRIPTION:
Women allocated to oxytocin only group will be given 10 units of oxytocin intramuscularly immediately after delivery of the fetus. Women allocated to the oxytocin plus uterine massage group will be will be given 10 units of oxytocin intramuscularly immediately after delivery of the fetus and will be provided with trans-abdominal uterine massage starting promptly after delivery of the fetus until delivery of the placenta. Collection of blood loss will be initiated immediately after delivery of the fetus by putting a drape under the woman's buttocks. Collected blood will be weighed and the amount will be recorded in grams.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old women delivering vaginally

Exclusion Criteria:

* women with bleeding disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Postpartum hemorrhage | during procedure
  The amount of blood loss after delivery of the fetus

SECONDARY OUTCOMES:
Duration of third stage of the labor | during procedure
  Delivery of the fetus and delivery of the placenta interval

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Kadirogullari P, Aslan Cetin B, Goksu M, Cetin Arslan H, Seckin KD. The effect of uterine massage after vaginal delivery on the duration of placental delivery and amount of postpartum hemorrhage. Arch Gynecol Obstet. 2024 Jun;309(6):2689-2695. doi: 10.1007/s00404-023-07211-5. Epub 2023 Sep 12. PMID 37698604